CLINICAL TRIAL: NCT03885466
Title: Nordic Walking for Individuals With Osteoporosis, Vertebral Fracture or Hyperkyphosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Royal University Hospital Foundation (Other); Saskatchewan Health Research Foundation (Other); Saskatchewan Centre for Patient-Oriented Research (Other)
Responsible Party: Principal Investigator, Saija Kontulainen, Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 140
Record Dates: First submitted 2019-02-21; First posted 2019-03-21 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Osteoporosis; Hyperkyphosis; Vertebral Fracture
Keywords: Nordic walking; Osteoporosis; Hyperkyphosis; Vertebral Fracture
MeSH Terms: conditions — Osteoporosis; Kyphosis; Spinal Fractures

STUDY DESIGN:
Intervention Model Description: A parallel group randomized control trial will be used to test our hypotheses. Participants randomized to the waiting-list control group will serve as controls for the baseline and 3-month measurements. The control group will receive the same 3-month Nordic walking intervention after their control follow-up measurements are completed.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research assistants and technicians collecting data will be blinded as to whether participants are in the exercise or control group. Participants will not be blinded for Nordic walking. All methods and reporting of the trial will follow Consolidated Standards of Reporting Trials (CONSORT) guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nordic walking (Experimental): Nordic walking exercise intervention, 3 times per week over 12 weeks
  Interventions: Behavioral: Nordic Walking exercise
- Control (No Intervention): Waiting list controls will be offered same Nordic walking intervention after 3 month follow-up measurements

INTERVENTIONS:
Behavioral: Nordic Walking exercise — Participants will initially train 3 times per week for 3 months. Training sessions will be led by trained peer- and/or student-instructors. Nordic walking sessions (starting at 20 and progressing to 60min/session) will include a warm-up, strengthening, and dynamic balance and stretching exercises in addition to Nordic walking, as per the Saskatoon Health Region guide (Saskatoon Health Region, 2014). Training (distance and intensity) will be progressive and individually set.
  Arms: Nordic walking

SUMMARY:
Nordic walking is currently offered by a number of health care practitioners as a form of exercise therapy for older adults at risk of fracture. These include older individuals with osteoporosis, previous vertebral fracture, or hyperkyphosis. To the investigators knowledge, this practice is not evidence-based and thus potentially problematic as benefits and safety of Nordic walking for individuals with osteoporosis, fractures, or hyperkyphosis are unknown. The proposed study will answer the following principal question: Does Nordic walking improve mobility, physical function, posture, and quality of life for ambulant community dwelling individuals who have osteoporosis, a history of osteoporotic fracture, or hyperkyphosis? Participants will be randomized into either the Nordic walking intervention group, or the waiting-list control group. Participants will initially train 3 times per week for 3 months, led by peer- and/or student-instructors. The Nordic walking training will depend on the participant's skill and comfort level and will consist of walking with poles over a distance set individually for each participant. The control group will receive the same 3-month Nordic walking intervention after their control follow-up measurements are completed.

DETAILED DESCRIPTION:
The investigators will include 160 individuals who have been diagnosed with osteoporosis, have history of osteoporotic fracture or hyperkyphosis (hunched-back posture). Participants will be randomized to either a Nordic walking intervention group or a waiting-list control group (the latter group will receive same intervention after the trial is completed). The pole-walking intervention will be 12 weeks in duration, including 3 weekly Nordic walking sessions (warm up, Nordic walking with posture and leg strengthening exercises and stretches) tailored to each participants. The investigators will define osteoporosis status at baseline (via DXA scans). The investigators will compare between group changes in dynamic balance, posture, quality of life, mobility, muscle strength, size and composition (using low radiation CT scans) after 3 months of Nordic walking intervention.

ELIGIBILITY:
Eligibility criteria for study participants:

* diagnosis of osteoporosis, past vertebral fracture or hyperkyphosis
* ambulatory (without the use of assistive devices)
* not currently involved in moderate-vigorous exercise training, including Nordic walking, more than once per week
* must not be diagnosed with Parkinson's disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Functional balance | 3-5 minutes
  Assessed by timed up and go test (TUG)
Quality of life score | 5-10 minutes
  Assessed by 36-Item Short Form Survey (SF-36). Survey consists of 36 questions with 8 sub-scales: Physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health. Responses range from 1-6 and are scored according to a key that values each answer from 0-100, where higher values are better outcomes. The average score of each sub-scale is recorded.
Kyphosis angle | 2-3 minutes
  Assessed using kyphometer

SECONDARY OUTCOMES:
Muscle strength | 2-4 minutes
  Assessed by sit-to-stand test
Mobility | 16-20 minutes
  Assessed by 6-minute walking test
Bone and muscle properties and estimated bone strength of the lower leg and forearm | 20-30 minutes
  Assessed by peripheral quantitative computed tomography (pQCT)
Total body lean tissue mass (g) | 10-20 minutes
  Assessed by dual-energy X-ray absorptiometry (DXA)
Proximal femur bone mineral density (g/cm^2) | 10-20 minutes
  Assessed by dual-energy X-ray absorptiometry (DXA)
Kyphosis angle | 3-5 minutes
  Assessed by flexicurve
Physical activity exercise confidence | 2-5 minutes
  Assessed by the Exercise self-efficacy scale. Scale consists of 10 questions with responses ranging from 1 (not confident at all) to 7 (very confident). Higher values are better outcomes. Sub-scale values are summed and total value is recorded.
Fear of falling | 2-5 minutes
  Assessed by the 10-item falls efficacy scale. Scale consists of 10 questions with responses ranging from 1 (not confident at all) to 10 (very confident). Higher values are better outcomes. Sub-scale values are summed and total value is recorded.
Physical activity | 7 days
  Recording minutes of physical activity using Actigraph wGT3X-BT accelerometer monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Saija Kontulainen, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website — https://research-groupstest.usask.ca/nws/index.php